CLINICAL TRIAL: NCT03958695
Title: A Randomized Clinical Trial Comparing a Tunable-tension Transobturator Tape (TTT) Versus Standard Transobturator Midurethral Tape (TOT) for the Surgical Treatment of Stress Urinary Incontinence in Women
Brief Title: A Tunable-tension Transobturator Tape vs Standard Transobturator Midurethral Tape for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Shkarupa Dmitry, Ph.D., Deputy Director for medical care, Chief Urologist of Saint Petersburg State University Clinic of advanced medical technologies n.a. N.I.Pirogov., Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTTvsTOT
Record Dates: First submitted 2019-05-05; First posted 2019-05-22 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Stress Urinary Incontinence
Keywords: midurethral sling; stress urinary incontinence; urinary incontinence; voiding dysfunction
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tunable-tension transobturator tape (TTT) (Active Comparator)
  Interventions: Device: Tunable-tension transobturator tape, Urosling-T (Lintex, LLC)
- Transobturator mid-urethral tape (TOT) (Active Comparator)
  Interventions: Device: Transobturator mid-urethral tape, Urosling (Lintex, LLC)

INTERVENTIONS:
Device: Tunable-tension transobturator tape, Urosling-T (Lintex, LLC) — A transobturator mid-urethral sling with the possibility of non-invasive tuning of its tension in the early postoperative period
  Arms: Tunable-tension transobturator tape (TTT)
Device: Transobturator mid-urethral tape, Urosling (Lintex, LLC) — A transobturator tension-free mid-urethral sling
  Arms: Transobturator mid-urethral tape (TOT)

SUMMARY:
This is the prospective randomized parallel groups trial with two participating centers (Department of Urology, Saint Petersburg State University Clinic of advanced medical technologies n.a. N.I.Pirogov, Saint Petersburg, Russia; Department of Urology, Regional Hospital №3, Chelyabinsk, Russia) designed to assess the efficacy and safety of tunable-tension transobturator tape and its ability to reduce the rate of postoperative voiding dysfunction comparing to standard transobturator midurethral sling.

DETAILED DESCRIPTION:
BACKGROUND A minimally invasive midurethral sling procedure is a favorite primary surgical method for the treatment of stress urinary incontinence (SUI). It is considered one of the most effective and safe anti-incontinence surgeries. The observed objective cure rate for transobturator sling is about 90%. However, this number may be wily because in most studies it does not exclude patients who achieved continence, but had voiding dysfunction. It is one of the most common complications of the midurethral sling, associated with the excess tape tension. The estimated rate of postoperative voiding dysfunction is up to 25%. There are few methods that allow to decrease tape tension after the surgery, such as urethral dilatation, sling mobilization, sling incision, complete excision of the tape and urethrolysis. All these methods are invasive, poorly controlled by the surgeon and are associated with the risk of recurrence of stress urinary incontinence.

PREOPERATIVE ASSESSMENT All patients who meet eligibility criteria will undergo a preoperative assessment: a detailed medical history, physical examination, vaginal examination, ICS-Uniform Cough Stress Test (ICS-UCST), uroflowmetry and ultrasound measurement of post-void residual volume (PVR). All patients will complete specific questionnaires, validated in Russia: Urogenital Distress Inventory 6 (UDI-6), International Conférence on Incontinence Questionnaire-Short Form (ICIQ-SF), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PICQ-12). The patients who will answer "Yes" to the question: "Do you experience urine leakage related to the feeling of urgency?" in UDI-6 questionnaire will undergo a urodynamic study to assess the presence and severity of detrusor overactivity.

MATERIALS AND METHODS The hypothesis is that TTT is non-inferior to TOT for SUI treatment. The sample size was calculated assuming an objective cure rate of 85% with TOT using a limit of equivalence of d=0,1 with 80% power. Thus 149 patients in each group are needed. We assume a drop-out rate of 30%, so in total 388 participants will be included in the study.

All enrolled patients will be randomly assigned to TTT or TOT treatment groups in equal ratio the day before the surgery, using computer randomization. The randomization will be performed by one resident urologist, who has no access to patients' data.

All surgical interventions will be performed by 4 urologists, performing at least 100 TOT surgeries per year. The next day after the surgery uroflowmetry values and PVR will be determined in all patients. In case of bladder outlet obstruction (BOO) symptoms, patients from TOT group will be recommended an intermittent self-catheterization for 6 weeks, or a urethral dilatation for choice. Patients from TTT group with BOO will undergo a procedure of non-invasive loosening of the tape under local anesthesia. The algorithm of uroflowmetry, PVR and tuning of the tape will be repeated until normal outflow values will be achieved. Also in patients from the TTT group, ICS-UCST will be estimated. If a patient will be experienced leakage a non-invasive tensioning of the tape under local anesthesia will be performed followed by uroflowmetry, PVR and additional tuning if necessary, until optimal tension will be achieved. The examination will be repeated on the day of discharge.

The postoperative assessment will be performed by 2 urologists, who will be blinded about the type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a woman with stress urinary incontinence or urodynamic mixed urinary incontinence with predominate SUI
* The subject is at least 18 years of age
* The subject has failed conservative treatment for at least 6 months
* The subject gave written consent to participate in the study,

Exclusion Criteria:

* The subject has an active urinary tract infection or skin infection in the region of surgery
* The subject has pelvic organ prolapse (POP) stage 2 or higher according to Pelvic Organ Prolapse Quantification system (POP-Q)
* The subject had prior surgery for SUI or POP
* The subject has predominate urge urinary incontinence
* The subject has a urogenital fistula, anatomical defect, stricture, diverticulum, new growth or any kind of abnormalities of the urethra
* The subject has chronic pelvic pain
* The subject has a system neurological disease, such as Parkinson's disease, Alzheimer disease and other dementias, multiple sclerosis, epilepsy etc
* The subject has pelvic cancer or the subject has undergone radiotherapy for treating pelvic cancer
* The subject has post void residual (PVR) >50 ml
* The subject has dysfunctional voiding and average flow rate (Qave) < 12 ml/s
* The subject is pregnant or disagrees to abstain from the pregnancy during the study
* The subject has any mental disorders affecting his ability to evaluate the risks of the treatment and make an independent decision on participation in the study
* The subject has an allergy on local anesthetics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Objective cure of stress urinary incontinence | 36 months (3 years)
  Objective cure is defined as the absence of urinary leakage during ICS-Uniform Cough Stress Test (ICS-UCST) in the absence of the bladder outlet obstruction

SECONDARY OUTCOMES:
Observed postoperative bladder outlet obstruction | Measured postoperatively at intervals of 1, 6, 12, 24 and 36 months postoperatively (3 years in total)
  Defined as average urine flow rate <12 ml/s or/and post void residual > 50 ml or/and urine retention
Subjective cure of stress urinary incontinence | Measured postoperatively at intervals of 1, 6, 12, 24 and 36 months postoperatively (3 years in total)
  Defined as an aswer "Never" to the question "Do you experience urine leakage related to physical activity, coughing or sneezing?" in UDI-6 questionnaire
Observed postoperative voiding dysfunction | Measured postoperatively at intervals of 1, 6, 12, 24 and 36 months postoperatively (3 years in total)
  Defined as the presence of any of the following complaints: slow urine stream, need to strain for voiding, intermittent stream, spraying, inability to void, incomplete bladder emptying, position-dependent voiding
Observed complications | Measured postoperatively at intervals of 1, 6, 12, 24 and 36 months postoperatively (3 years in total)
  Presense of any adverse effects such as: bleeding, haematoma, organ perforation, wound infection, urinary tract infection, pelvic pain, mesh extrusion in the vagina, mesh erosion into the urinary tract, dyspareunia de novo, de novo urgency
The assessment of the impact of treatment on the quality of life: Urogenital Distress Inventory (UDI-6) questionnaire | Measured postoperatively at intervals of 12, 24 and 36 months postoperatively (3 years in total)
  Measured through the Urogenital Distress Inventory (UDI-6) questionnaire, validated in Russia. The score varies from 0 to 100. The basic interpretation of the score is that the higher the score, the worse the outcome.
The assessment of self-reported success of the treatment | Measured postoperatively at intervals of 12, 24 and 36 months postoperatively (3 years in total)
  Measured through the International Conférence on Incontinence Questionnaire Short Form (ICIQ-SF) questionnaire, validated in Russia. The questionnaire is a subjective measure of severity of urinary loss and patients' quality of life. The score varies from 0 to 21. The higher the score indicates greater severity of urinary incontinence: 1-5 - slight, 6-12 - moderate, 13-18 - severe, 19-21 - very severe.
The assessment of the impact of treatment on sexual function | Measured postoperatively at intervals of 12, 24 and 36 months postoperatively (3 years in total)
  Measured through the scoring of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) validated in Russia. The scale evaluates sexual function in patients with urinary incontinence and/or POP. The responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Items 1 - 4 are reversely scored and a total of 48 is the maximum score. The higher scores indicate better sexual function. Up to two missing responses are accepted. The total score sum with missing values is calculated by multiplying the number of items by the mean of the responses to the items reported by that person.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shkarupa, PhD, MD, Principal Investigator — Saint Petersburg State University, Russia
Locations (2):
- Russia (2):
  - Regional Clinic Hospital №3, Chelyabinsk
  - Saint Petersburg State University Clinic of advanced medical technologies n.a. N.I.Pirogov, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No